CLINICAL TRIAL: NCT02477657
Title: Palliative Care Outcomes in the Management of Malignant Ascites by Interventional Radiology
Status: Withdrawn | Type: Observational
Why Stopped: Industry funding not received. No subjects enrolled.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 26813
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Refractory Malignant Ascites
Keywords: Adult patients with refractory malignant ascites secondary to GU or GI malignancy.
MeSH Terms: interventions — Paracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Paracentesis — Paracentesis
Device: Tunneled Intraperitoneal Drain (IPD) — Tunneled Intraperitoneal Drain (IPD)
Device: Peritoneal-Venous shunts (PVS) — Peritoneal-Venous shunts (PVS)

SUMMARY:
Malignant ascites leads to significant morbidity in patients with terminal cancer. Paracentesis can provide relief, but repeat hospital visits, pain, and short duration of relief after paracentesis are detrimental to quality of life(QOL). Two devices are available as alternatives to paracentesis. The impact of either device on QOL has not fully been explored. A pilot nonrandomized trial measuring palliative care QOL and ascites symptom relief using validated survey instruments is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Refractory malignant ascites defined as ascites requiring more than one paracentesis to control patient symptoms despite medical therapy with diuretics and a. peritoneal fluid with cytology positive for malignant cells OR
* Known malignancy with imaging findings of peritoneal carcinomatosis .
* Eastern Cooperative Oncology Group (ECOG) performance score 3
* Age greater than or equal to 18
* Capable of giving informed consent

Exclusion Criteria:

* Life expectancy less than one month
* Coagulopathy defined as international normalized ration (INR) >2 which cannot be corrected with fresh frozen plasma
* Platelet count <50,000/microliter, which cannot be corrected with platelet transfusion
* Active skin infections at sites where PVS would be inserted
* Presence of infectious peritonitis or bacteremia
* Neutropenia
* American Heart Association Class D congestive heart failure (ie New York Heart Association Class IV)
* Stage 5 CKD (ie GFR < 15 mL/min)
* Severe hypoalbuminemia defined as < 2.2 g/dL
* Loculated or hemorrhagic ascites
* History of bleeding gastroesophageal varices
* Inability to provide informed consent
* Unable to participate in neuropsychological tests / questionnaires
* Pregnant or nursing women
* Anasarca

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with refractory malignant ascites secondary to GU or GI malignancy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Nadolski, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States